CLINICAL TRIAL: NCT05670405
Title: The Trauma PORTAL Project: A Randomized Controlled Trial of a Virtual Asynchronous Psychoeducational Psychotherapy Treatment for Survivors of Childhood Interpersonal Trauma
Brief Title: The Trauma PORTAL Project: a Virtual Asynchronous Treatment for Interpersonal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Dana Ross, Psychiatrist, Trauma Therapy Program, Women's College Hospital, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0083-E
Record Dates: First submitted 2022-11-30; First posted 2023-01-04 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Psychological Trauma
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma PORTAL Intervention (Experimental): The treatment group will complete the Trauma PORTAL intervention in 9 weeks. The participants will be asked to complete clinical measures at baseline, 8 weeks, and 16 weeks.
  Interventions: Other: The Trauma PORTAL
- Care-as-Usual (No Intervention): The control group will receive care-as-usual, remaining on the waitlist for the regular TTP R&R groups. Participants in the CUC group will be asked to complete clinical measures at time points corresponding to the ITC group's baseline (prior to starting week one) and post-intervention (i.e. primary endpoint, end of week 8). Both groups will complete the clinical measures eight weeks later (16-week time point).

INTERVENTIONS:
Other: The Trauma PORTAL — Participants will have 9 weeks to complete the 8 modules which each take on average 45 minutes to complete. Each module consists of psychoeducational handouts, videos, interactive exercises, and discussion topics that has been adapted from the R&R curriculum. The participants will also receive a pdf of the handouts from the modules, which can be used to take notes or refer back to in the future.
  There will be an optional 60-minute weekly virtual group session for participants to engage with other participants in their group and for group facilitator providers to discuss the materials covered and answer any questions. Participants will join a Zoom video group visit to access the group. Each weekly group will be facilitated by 2 clinicians specializing in trauma-focused therapy within the WCH TTP who have extensive experience with in-person and virtual synchronous R&R.
  Arms: Trauma PORTAL Intervention

SUMMARY:
Virtual delivery of mental health care is an emerging strategy for increasing access and enhancing the delivery of mental health services; however, evidence that virtual interventions are an efficacious form of therapy is limited. An asynchronous virtual treatment program that allows patients to access program material at any time could be a widely accessible, cost-effective alternative to in-person or synchronous virtual group therapy. The Trauma Therapy Program (TTP) at Women's College Hospital (WCH) follows clinical guidelines for the treatment of complex post-traumatic stress disorder that recommend a staged approach to treatment for adults suffering from the sequelae of childhood interpersonal trauma (CIT). The initial stage is safety and stabilization; in TTP, this begins with the Resourced and Resilient (R&R) group, a stage 1 trauma-focused psychoeducational psychotherapy group. Psychoeducational psychotherapy is a widely used approach to help patients understand the impact of trauma, challenge maladaptive behaviour patterns, learn safer coping skills and reduce trauma-related symptoms as part of a comprehensive approach to the treatment of PTSD. To address gaps in equitable access to trauma-focused care, the investigators developed the Trauma PORTAL: Providing Online tRauma Therapy using an Asynchronous Learning platform. The investigators developed an asynchronous virtual multimedia version of R&R consisting of 8 modules, called the Trauma PORTAL; previously called electronic Resourced and Resilient or e-R&R. The investigators then conducted an open-label pilot study where the Trauma PORTAL intervention was offered that included access to the asynchronous virtual modules, along with an optional weekly 1-hour synchronous virtual group that offers patients an opportunity to ask questions about content from the modules. Preliminary data from the investigators' open-label eR&R pilot study demonstrates feasibility, usability, and acceptability, as well as a significant improvement in PTSD symptoms from pre- to post-group. This phase of the Trauma PORTAL project seeks to test the efficacy and further assess the intervention processes, including recruitment, retention, acceptability, and adherence to the Trauma PORTAL intervention through a randomized controlled trial.

DETAILED DESCRIPTION:
The investigators aim to conduct a randomized controlled trial to determine the efficacy of the Trauma PORTAL intervention. The Trauma PORTAL is an asynchronous virtual multimedia version of the stage 1 trauma-focused psychoeducational psychotherapy group called Resourced & Resilient (R&R) in the Trauma Therapy Program (TTP) at Women's College Hospital (WCH). The TTP is a specialized trauma-focused therapy service for persons with childhood histories of trauma. The program offers confidential, time-limited and primarily group-based psychotherapy to adults who have experienced childhood interpersonal trauma, including physical, sexual, and emotional abuse and/or neglect that occurred between the ages of 0-18. The TTP comprises an interdisciplinary team of trauma therapists with backgrounds in psychiatry, psychotherapy, psychology, social work, and nursing.

The Trauma PORTAL intervention consists of 8 online modules that participants can complete at the participants own pace, with optional once-weekly "live" virtual sessions facilitated by trauma therapists in the TTP. The investigators specifically aim to measure clinical symptoms to generate estimates of the effect of the Trauma PORTAL intervention on clinical measures of PTSD, depression, anxiety, and emotion regulation compared to a care-as-usual condition. The investigators will also evaluate the intervention processes, including recruitment, retention, acceptability and adherence to inform spread and scale post-trial if the intervention is demonstrated to be effective.

Individuals will be recruited from the waitlist for the "live" synchronous virtual or in-person R&R group in the TTP.

Individuals will be randomized to receive the Trauma PORTAL intervention (immediate treatment condition, ITC) or treatment as usual while on a waitlist (care-as-usual condition, CUC). Participants randomized to CUC will remain on the waitlist for live R&R and complete clinical measures at the same time points as the ITC group. All participants will complete clinical measures at baseline, 8 weeks, and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old; and
* Self-report childhood interpersonal trauma (physical, sexual, emotional, neglect) prior to age 18; and
* A diagnosis of PTSD aligned with the Mini International Neuropsychiatric Interview Module H; and
* Access to appropriate device and internet connection to access the intervention; and
* Attended an orientation session for the Trauma Therapy Program at WCH; and
* Suitable for Trauma PORTAL intervention (confirmed by clinical assessment with a TTP Therapist)*

  * Participants will not be included if, based on a clinical assessment with a TTP therapist, there is a concern that the participant has: (1) significant difficulty with self-regulation which make them unsuitable for an outpatient asynchronous intervention, (2) cognitive impairments that would impede understanding and processing of educational material, (3) significant case management needs that would result in lack of suitability for asynchronous online group therapy, or (4) for any other clinical reason, at the discretion of the assessing TTP therapist.

Exclusion Criteria:

* Have had active alcohol or substance use disorder in the past 3 months; or
* Have active symptoms of mania or psychosis, or active suicidal ideation; or
* Have had psychiatric hospitalization in the past 6 months; or
* Are unable to complete study procedures in English (intervention not yet translated)
* Previously completed an R&R group with an approved provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5) score | At baseline, week 8 and week 16
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The self-report rating scale is 0-4 for each symptom. The min and max values are 0 and 80, with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Change in Clinician-Administered Post-Traumatic Stress Disorder Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Past Month score (CAPS-5 Past Month) score | At baseline, week 8 and week 16
  The CAPS-5 - Past Month score is a 30-item structured interview that can be used to make a current (past month) or lifetime diagnosis of PTSD and assess PTSD symptoms over the past week. The min and max values are 0 to 80, with higher scores indicating worse outcome.
Change in Difficulties in Emotion Regulation Scale (DERS-18) score | At baseline, week 8 and week 16
  The DERS-18 is a multi-dimensional assessment of emotion regulation and dysregulation. It consists of a self-reported 18-item questionnaire that assesses 6 subscales: lack of awareness of one's emotions, lack of clarity about the nature of one's emotions, lack of acceptance of one's emotions, lack of access to effective emotion regulation strategies, lack of ability to engage in goal-directed activities during negative emotions, and lack of ability to manage one's impulses during negative emotions. Each subscale consists of 3 items, which are rated on a scale of 1 (almost never) to 5 (almost always). The min and max values are 18 and 90, with higher scores indicating worse outcome.
Change in Short Self-Compassion Scale (Short SCS) score | At baseline, week 8 and week 16
  The Short SCS is a 12-item survey assessing 6 subscales: self-judgement, self-kindness, common humanity, isolation, mindfulness, and overidentification. Questions are rated on a 5-point scale ranging from 1 (almost never) to 5 (almost always) with subscale scores computed by calculating the mean of subscale item responses. The min and max values are 12 and 60, with higher scores indicating greater self-compassion.

OTHER OUTCOMES:
Change in Health Service Utilization Questionnaire responses | At baseline and week 16
  The Health Service Utilization Questionnaire will ask for Information on participant mental health service use to to capture any changes that could affect outcomes over the course of the Trauma PORTAL intervention. Increased health service utilization may indicate a worse outcome.
General Internet Attitude Scale | Baseline
  The General Internet Attitude Scale is a validated baseline questionnaire measuring the participants beliefs and attitudes about using the Internet. The 21 items assess four subscales: Social benefit, Negative affect, Exhilaration, and Detriment. Questions are rated on a 5-point scale (strongly disagree, slightly disagree, no opinion, slightly agree, agree). Higher scores indicate more positive attitudes toward the internet. This scale will provide valuable information regarding study participants' levels of comfort with the Internet, which will likely affect acceptance of an eHealth intervention such as the Trauma Portal intervention by participants.
Health Service Research Question Measures - Recruitment Data | Through study completion, an average of 1 year
  The research team will collect recruitment numbers and rate, and reasons for ineligibility and non-consent; and the number of days required to fill each "participant group" (i.e. up to 25 participants)
Health Service Research Question Measures - Adherence Data | Through study completion, an average of 1 year
  Adherence data will be collected looking at rates of weekly login and module completion, as well as overall Trauma PORTAL completion, Number of weekly live synchronous groups attended, Length of time spent on weekly modules, Reasons for non-use or discontinuation of the intervention, and completion of baseline and post-intervention measures
Health Service Research Question Measures - Safety Data | Through study completion, an average of 1 year
  Safety data will be collected including the number of safety concerns, the need for trial psychiatrist to assess and/or assume care of the participant, and adverse events (i.e. participants meeting stopping criteria)
Health Service Research Question Measures - Healthy System Implications Data | Through study completion, an average of 1 year
  Health system implications will be evaluated by conducting a clinical chart review to identify the number of weekly online group sessions attended, if any additional contacts were required throughout the course of the intervention, and results of the assessment for next steps.
Acceptability of intervention in the target population | At week 8
  After completion of the Trauma PORTAL intervention, treatment group participants will be asked to complete an Intervention Acceptability Questionnaire comprised of open and closed ended questions. Closed ended questions will elicit feedback on (1) usability of the Trauma PORTAL; (2) benefits of the Trauma PORTAL intervention including usefulness and increased accessibility of healthcare; (3) perceived security of personal health information; (4) concerns regarding continuity of care; and (5) overall user satisfaction.
Iterative Feedback Form | Once weekly for 8 weeks
  Every week a short but optional Iterative Feedback Form (IFF) will be sent to the treatment group participants. These forms will be reviewed by the research team on a weekly basis. There will be questions for participants to let us know how long they spent on each module, and reasons for not completing it (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Dana C. Ross, MD, MSc, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada